CLINICAL TRIAL: NCT00945672
Title: A PHASE 2 DOUBLE-BLINDED, RANDOMIZED, PLACEBO-CONTROLLED, MULTICENTER STUDY EVALUATING THE SAFETY, TOLERABILITY AND PHARMACOKINETICS/ PHARMACODYNAMICS OF PF-04360365 IN MILD TO MODERATE ALZHEIMER'S DISEASE PATIENTS
Brief Title: A Multiple Dose Study of PF-04360365 In Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: A9951007; 2009-011172-30 (EudraCT Number); PIB/PET IMAGING (Other: Alias Study Number)
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease amyloid imaging antibody
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PF-04360365 10 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 10 mg/kg
- PF-04360365 7.5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 7.5 mg/kg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: PF-04360365 10 mg/kg — 10 mg/kg every 90 days (5 total doses)
  Arms: PF-04360365 10 mg/kg
Biological: PF-04360365 7.5 mg/kg — 10 mg/kg loading dose followed by 7.5 mg/kg monthly maintenance dosing (total of 13 doses)
  Arms: PF-04360365 7.5 mg/kg
Drug: placebo — placebo administered every 90 days or monthly to match experimental treatment arms.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether multiple dose administration is safe and well tolerated in patients with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non childbearing potential, age > or = 50.
* Diagnosis of probable Alzheimer's disease, consistent with criteria from both:

  * National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA).
  * Diagnostic and Statistical Manual of Mental Disorders (DSM IV).
* Mini-mental status exam score of 16-26 inclusive.
* Rosen-Modified Hachinski Ischemia Score of < or = 4.

Exclusion Criteria:

* Diagnosis or history of other demential or neurodegenerative disorders.
* Diagnosis or history of clinically significant cerebrovascular disease.
* Specific findings on magnetic resonance imaging (MRI); cortical infarct, micro hemorrhage, multiple white matter lacunes, extensive white matter abnormalities.
* History of autoimmune disorders.
* History of allergic or anaphylactic reactions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08-06 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2011-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Sweden (4):
  - Sahlgrenska Sjukhuset, CTC, Gothenburg
  - Malmo Sjukhus, Neuropsykiatriska Kliniken, Malmo
  - Sahlgrenska Universitetssjukhuset, Minnesmottagningen, Mölndal
  - Karolinska Universitetssjukhuset Huddinge, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951007&StudyName=A%20Multiple%20Dose%20Study%20of%20PF-04360365%20In%20Patients%20With%20Mild%20to%20Moderate%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04360365 10 mg/kg (Cohort Q): Participants received PF-04360365 10 milligram per kilogram (mg/kg) intravenous infusion over 10 minutes on Day 1 and then once in every 3 months up to a maximum duration of 12 months.
- Placebo (Cohort Q): Participants received placebo matched to PF-04360365 10 mg/kg intravenous infusion over 10 minutes on Day 1 and then once in every 3 months up to a maximum duration of 12 months.
- PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M): Participants received PF-04360365 loading dose of 10 mg/kg intravenous infusion over 10 minutes on Day 1, followed by PF-04360365 7.5 mg/kg intravenous infusion over 10 minutes every month starting from Month 1 up to 12 months.
- Placebo (Cohort M): Participants received placebo matched to PF-04360365 on Day 1, followed by placebo intravenous infusion over 10 minutes every month starting from Month 1 up to 12 months.
Period: Overall Study
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Started | 12 | 6 | 12 | 6
Completed | 12 | 6 | 12 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 infusion of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M) | Total
Number analyzed (Participants) | 12 | 6 | 12 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.4) | 71.3 (8.5) | 69.8 (7.5) | 65.8 (8.3) | 67.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 5 | 15
  Male | 8 | 3 | 9 | 1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to 6 months after last dose (up to 18 months) that were absent before treatment or worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Day 1 up to 6 months after last dose of study medication (up to 18 months)
Population: Safety analysis set included all randomized participants who received at least 1 infusion of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
Participants
  AEs | 9 | 5 | 10 | 5
  SAEs | 2 | 1 | 1 | 0

2. Primary Outcome: Number of Participants With Change From Baseline in Brain Magnetic Resonance Imaging (MRI) Abnormalities
Description: Number of participants with new clinical findings not evident on the baseline scans, such as brain edema, hemorrhage, encephalitis and other pathology (cerebral edema, cerebral/meningeal enhancement, micro hemorrhage, parenchymal hematoma, subarachnoid hemorrhage, subdural hematoma, cortical infarcts, subcortical grey matter infarcts, white matter infarcts and white matter hyper intensities) were assessed from structural magnetic resonance imaging (MRI). Participants with brain abnormality other than those listed above assessed using MRI scan were reported under 'other' category. Only those MRI findings in which at least 1 participant had event, were reported.
Time Frame: Baseline up to Month 18
Population: Safety analysis set included all randomized participants who received at least 1 infusion of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
Participants
  Micro Hemorrhage | 1 | 0 | 1 | 1
  Other | 2 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Gadolinium Use in Brain Magnetic Resonance Imaging (MRI)
Description: Brain MRI included gadolinium contrast if investigator determined this was necessary for participant care either based on clinical signs or the non-contrast MRI. This decision was made by the investigator on the basis of change in the clinical examination or in response to a possible abnormality seen on the non-contrast brain MRI.
Time Frame: Baseline up to Month 18
Population: Safety analysis set included all randomized participants who received at least 1 infusion of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Change From Baseline in Amyloid Load at Month 13 Using Positron Emission Tomography (PET) Technique: Cohort M
Description: Quantitative amyloid imaging was performed using PET technique using [11C] Pittsburgh Compound B (PIB) for following brain areas: frontal, temporal, parietal and occipital cortices, anterior and posterior cingular cortex, cerebellum, pons, and subcortical white matter. For target regions of interest, beta-amyloid plaque imaging radiotracer (PIB) retention data was expressed as standard uptake value ratio (SUVR) which was defined as a ratio of radioactivity uptake of the target region relative to the cerebellum reference region. This outcome measure was planned to be analyzed only for cohort M.
Time Frame: Baseline, Month 13
Population: Per Protocol (PP) analysis set included all participants who had received the study drug infusions consistent with the protocol specified procedures, had successful PET scans at Month 13, and had no major protocol deviations. Only participants in cohort M were planned to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Standard update value ratio
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6
Standard update value ratio
  Baseline: Frontal Cortex | 2.781 (0.6769) | 2.835 (0.3775)
  Baseline: Parietal Cortex | 2.480 (0.5175) | 2.647 (0.4020)
  Baseline: Lateral Temporal Cortex | 2.492 (0.4945) | 2.626 (0.3327)
  Baseline: Occipital Cortex | 2.085 (0.4064) | 1.994 (0.2066)
  Baseline: Cerebellum | 1.000 (0.0000) | 1.000 (0.0000)
  Baseline: Striatum | 2.325 (0.4351) | 2.440 (0.3468)
  Baseline: Anterior Cingulum | 2.723 (0.6085) | 2.845 (0.3109)
  Baseline: Temporal Medial | 1.557 (0.1693) | 1.615 (0.1334)
  Baseline: Posterior Cingulum | 2.866 (0.5547) | 2.927 (0.3624)
  Baseline: Pons | 2.042 (0.3195) | 2.091 (0.3871)
  Baseline: Subcortical White Matter | 2.315 (0.3442) | 2.407 (0.3180)
  Change at Month 13: Frontal Cortex | -0.092 (0.3081) | -0.096 (0.3243)
  Change at Month 13: Parietal Cortex | -0.030 (0.2039) | -0.113 (0.3309)
  Change at Month 13: Lateral Temporal Cortex | -0.056 (0.2485) | -0.094 (0.2956)
  Change at Month 13: Occipital Cortex | -0.066 (0.2027) | 0.047 (0.2409)
  Change at Month 13: Cerebellum | 0.000 (0.0000) | 0.000 (0.0000)
  Change at Month 13: Striatum | -0.047 (0.1602) | -0.091 (0.2568)
  Change at Month 13: Anterior Cingulum | -0.103 (0.2397) | -0.068 (0.3245)
  Change at Month 13: Temporal Medial | -0.009 (0.0960) | -0.025 (0.2255)
  Change at Month 13: Posterior Cingulum | -0.065 (0.2770) | -0.103 (0.3539)
  Change at Month 13: Pons | -0.026 (0.2034) | -0.013 (0.2181)
  Change at Month 13: Subcortical White Matter | -0.083 (0.2047) | -0.024 (0.2781)

5. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of PF-04360365 at 0 Hour on Day 0
Description: Samples for PF-04360365 concentration were assayed using a validated, sensitive and specific enzyme-linked immunosorbent assay method.
Time Frame: 0 hour on Day 0 (Day prior to dosing)
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure. Only participants receiving PF-04360365 were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11 | 12
Nanogram per milliliter (ng/mL) | 0.00 (0.00) | 0.00 (0.00)

6. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 1
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 1
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure. Only participants receiving PF-04360365 were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12 | 11
ng/mL | 0.00 (0.00) | 0.00 (0.00)

7. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 1
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11 | 12
ng/mL | 191080.73 (27645.17) | 190826.33 (64016.37)

8. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 10: Cohort M
Description: as for outcome 5
Time Frame: 216 hours post dose on Day 1 (samples taken on Day 10)
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure. Only participants receiving PF-04360365 every month (cohort M) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 4
ng/mL
  CSF | 167.25 (52.68)
  Plasma | 77466.25 (11446.87)

9. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 20: Cohort M
Description: as for outcome 5
Time Frame: 456 hours post dose on Day 1 (samples taken on Day 20)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 4
ng/mL
  CSF | 192.50 (90.50)
  Plasma | 68219.25 (18837.66)

10. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 at 0 Hour on Day 30: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 30
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure and 'Number Analyzed' signifies participants evaluable for the specified rows. Only participants receiving PF-04360365 every month (cohort M) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11
ng/mL
  CSF: number analyzed (Participants) | 4
  CSF | 185.33 (86.53)
  Plasma | 46321.00 (5902.85)

11. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 30: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11
ng/mL | 196752.82 (25216.35)

12. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 40: Cohort Q
Description: as for outcome 5
Time Frame: 936 hours post dose on Day 1 (samples taken on Day 40)
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure. Only participants receiving PF-04360365 every 3 months (cohort Q) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q)
Number analyzed (Participants) | 4
ng/mL
  CSF | 121.73 (35.25)
  Plasma | 34794.50 (4381.87)

13. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 50: Cohort Q
Description: as for outcome 5
Time Frame: 1176 hours post dose on Day 1 (samples taken on Day 50)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q)
Number analyzed (Participants) | 4
ng/mL
  CSF | 107.03 (44.93)
  Plasma | 40038.50 (11862.03)

14. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 60: Cohort Q
Description: as for outcome 5
Time Frame: 1416 hours post-dose on Day 1 (samples taken on Day 60)
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure and 'Number Analyzed' signifies participants evaluable for the specified rows. Only participants receiving PF-04360365 every 3 months (cohort Q) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q)
Number analyzed (Participants) | 4
ng/mL
  CSF | 84.50 (25.51)
  Plasma: number analyzed (Participants) | 3
  Plasma | 22917.00 (4432.31)

15. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hours on Day 60: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 60
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Only participants receiving PF-04360365 every month (cohort M) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 62261.92 (13196.38)

16. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 60: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 60
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 10
ng/mL | 199861.90 (33651.83)

17. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 at 0 Hour on Day 90
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 90
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here 'Number Analyzed' signifies participants evaluable for specified row for each treatment arm, respectively. Only participants receiving PF-04360365 were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12 | 12
ng/mL
  CSF: number analyzed (Participants) | 4 | 0
  CSF | 61.15 (11.76) |
  Plasma | 16094.08 (4932.12) | 68110.83 (12594.63)

18. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 90
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11 | 10
ng/mL | 218031.73 (30864.41) | 212299.30 (20405.36)

19. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 120: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 120
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 73285.25 (20795.73)

20. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 120: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 10
ng/mL | 227156.80 (23587.30)

21. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 150: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 150
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 76083.50 (19076.47)

22. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 150: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 150
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11
ng/mL | 222737.91 (28714.06)

23. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 at 0 Hour on Day 180
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 180
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here 'Number Analyzed' signifies participants evaluable for specified rows for each treatment arm, respectively. Only participants receiving PF-04360365 were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12 | 12
ng/mL
  CSF: number analyzed (Participants) | 8 | 11
  CSF | 89.20 (26.12) | 324.82 (119.92)
  Plasma | 23708.42 (5039.46) | 76593.58 (14452.02)

24. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 180
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 180
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11 | 10
ng/mL | 226842.91 (22478.66) | 210905.00 (26474.96)

25. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 210: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 210
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 77315.33 (14237.02)

26. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 210: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 210
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 223667.00 (28942.32)

27. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 240: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 240
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 82563.83 (21690.43)

28. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 240: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 240
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11
ng/mL | 223715.91 (29306.75)

29. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 270
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 270
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11 | 12
ng/mL | 22140.00 (8996.92) | 69838.25 (16735.16)

30. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 270
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 270
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 7 | 11
ng/mL | 219643.86 (21122.06) | 218116.27 (20328.81)

31. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 300: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 300
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11
ng/mL | 71822.18 (16913.55)

32. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 300: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 300
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 10
ng/mL | 227333.20 (30922.55)

33. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 330: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 330
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 71668.67 (19448.75)

34. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 330: Cohort M
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 330
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 9
ng/mL | 216841.22 (38575.76)

35. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 at 0 Hour on Day 360
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 360
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Only participants receiving PF-04360365 were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12 | 12
ng/mL
  CSF | 68.71 (27.52) | 240.19 (93.38)
  Plasma | 20347.00 (8570.57) | 70238.33 (23030.37)

36. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0.25 Hours on Day 360
Description: as for outcome 5
Time Frame: 0.25 hours post-infusion start on Day 360
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 11 | 11
ng/mL | 222927.73 (29419.72) | 213278.09 (31361.98)

37. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 720 Hours Post-dose on Day 360: Cohort Q
Description: as for outcome 5
Time Frame: 720 hours post-dose on Day 360 (samples taken on Day 390)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q)
Number analyzed (Participants) | 9
ng/mL | 59095.22 (9470.32)

38. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 390: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 390
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure. Only participants receiving PF-04360365 every month (cohort M) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 74846.08 (25913.06)

39. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hours on Day 540: Cohort Q
Description: as for outcome 5
Time Frame: 0 hours (pre-dose) on Day 540
Population: PK analysis set included all participants who received at least 1 infusion of PF-04360365. Only participants receiving PF-04360365 every 3 months (cohort Q) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q)
Number analyzed (Participants) | 12
ng/mL | 6245.83 (3567.48)

40. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 540: Cohort M
Description: as for outcome 5
Time Frame: 0 hour (pre-dose) on Day 540
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12
ng/mL | 5987.08 (3571.64)

41. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 0 Hour on Day 0
Description: A-beta is a peptide fragment of the amyloid precursor protein (found in the brain of participants suffering from of Alzheimer's disease (AD). In this outcome, CSF concentration of 3 variants of A-beta were reported: A-beta (1-X), A-beta (1-40) and A-beta (1-42).
Time Frame: 0 hour on Day 0 (Day prior to dosing)
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 infusion of study medication.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/mL)
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
Picogram per milliliter (pg/mL)
  A-beta 1-x | 31150.00 (9063.66) | 28533.33 (5269.41) | 30497.50 (16885.00) | 28500.00 (8696.44)
  A-beta 1-40 | 15794.17 (7569.38) | 13296.67 (2428.35) | 11688.33 (3813.40) | 12215.00 (2674.13)
  A-beta 1-42 | 1003.75 (358.30) | 882.00 (185.95) | 758.67 (204.65) | 870.00 (270.25)

42. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 216 Hours Post-dose on Day 1: Cohort M
Time Frame: 216 hours post-dose on Day 1
Population: FAS included all randomized participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure. Only participants receiving PF-04360365 or placebo every month (cohort M) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 4 | 1
pg/mL
  A-beta 1-x | 22.32 (17.55) | -21.21 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  A-beta 1-40 | 9.24 (44.06) | 1.43 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  A-beta 1-42 | -0.46 (14.59) | -3.78 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.

43. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 456 Hours Post-dose on Day 1: Cohort M
Time Frame: 456 hours post-dose on Day 1
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 4 | 1
pg/mL
  A-beta 1-x | -2.38 (14.01) | -5.95 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  A-beta 1-40 | 4.23 (25.16) | -8.75 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  A-beta 1-42 | 8.14 (31.37) | -24.57 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.

44. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 0 Hour on Day 30: Cohort M
Time Frame: 0 hour (pre-dose) on Day 30
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 4 | 2
pg/mL
  A-beta 1-x | 0.80 (31.57) | -0.79 (30.68)
  A-beta 1-40 | 43.33 (20.67) | -17.07 (19.05)
  A-beta 1-42 | 14.15 (17.45) | -13.98 (12.48)

45. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 936 Hours Post-dose on Day 1: Cohort Q
Time Frame: 936 hours post-dose on Day 1 (Samples taken on Day 40)
Population: FAS included all randomized participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure. Only participants receiving PF-04360365 or placebo every 3 months (cohort Q) were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q)
Number analyzed (Participants) | 4 | 2
pg/mL
  A-beta 1-x | 16.78 (9.69) | 5.05 (3.71)
  A-beta 1-40 | 26.77 (16.01) | 160.62 (51.13)
  A-beta 1-42 | 17.30 (14.03) | -7.40 (13.74)

46. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 1176 Hours Post-dose on Day 1: Cohort Q
Time Frame: 1176 hours post-dose on Day 1 (Samples taken on Day 50)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q)
Number analyzed (Participants) | 4 | 2
pg/mL
  A-beta 1-x | 12.35 (11.45) | -1.60 (9.02)
  A-beta 1-40 | -17.98 (37.02) | -6.67 (9.43)
  A-beta 1-42 | 2.32 (16.51) | -3.36 (18.68)

47. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 1416 Hours Post-dose on Day 1: Cohort Q
Time Frame: 1416 hours post-dose on Day 1 (Samples taken on Day 60)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q)
Number analyzed (Participants) | 4 | 2
pg/mL
  A-beta 1-x | 9.62 (6.51) | 0.04 (1.33)
  A-beta 1-40 | 27.85 (35.55) | -5.61 (0.44)
  A-beta 1-42 | 9.52 (14.31) | -12.08 (2.95)

48. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 0 Hour on Day 90: Cohort Q
Time Frame: 0 hour (pre-dose) on Day 90
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q)
Number analyzed (Participants) | 4 | 1
pg/mL
  A-beta 1-x | -0.51 (8.96) | -15.57 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  A-beta 1-40 | 27.67 (40.65) | -23.23 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  A-beta 1-42 | -15.62 (18.01) | -38.65 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.

49. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 0 Hour on Day 180
Time Frame: 0 hour (pre-dose) on Day 180
Population: FAS included all randomized participants who received at least 1 infusion of PF-04360365. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this measure and 'Number Analyzed' signifies participants evaluable for specified amyloid beta for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 8 | 4 | 12 | 5
pg/mL
  A-beta 1-x | -37.94 (9.81) | -44.49 (10.99) | 13.91 (21.25) | -0.57 (23.16)
  A-beta 1-40 | -60.93 (13.99) | -60.42 (7.98) | 179.14 (121.44) | 147.17 (126.47)
  A-beta 1-42: number analyzed (Participants) | 7 | 4 | 12 | 5
  A-beta 1-42 | 18.57 (19.99) | -4.18 (22.66) | 75.58 (45.47) | -15.77 (34.09)

50. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (A-beta 1-x), Amyloid Beta 1-40 (A-beta 1-40) and Amyloid Beta 1-42 (A-beta 1-42) at 0 Hour on Day 360
Time Frame: 0 hour (pre-dose) on Day 360
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 5 | 12 | 5
pg/mL
  A-beta 1-x | -16.70 (22.23) | -30.01 (11.85) | -27.69 (28.11) | -42.16 (17.77)
  A-beta 1-40: number analyzed (Participants) | 9 | 4 | 12 | 5
  A-beta 1-40 | 98.33 (133.77) | 35.60 (122.29) | 3.07 (69.15) | 56.66 (90.93)
  A-beta 1-42: number analyzed (Participants) | 12 | 4 | 12 | 5
  A-beta 1-42 | -26.70 (40.32) | -40.24 (14.77) | 49.15 (54.18) | -27.46 (11.27)

51. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) Total Score at Months 3, 6, 9, 13 and 18
Description: ADAS-cog is a structured scale assessing the severity of cognitive impairment in Alzheimer's Disease. It comprises of following 11 items (range): word recall (0-10), naming objects and fingers (0-5), following commands (0-5), constructional praxis (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), recall of test instructions (0-5), spoken language ability (0-5), word-finding difficulty (0-5), comprehension of spoken language (0-5). The total score was calculated as the sum of the scores for the 11 items. ADAS-cog total score ranges from 0 (no impairment) to 70 (maximum impairment). Higher total and individual item scores indicate greater cognitive impairment.
Time Frame: Baseline, Month 3, 6, 9, 13, 18
Population: FAS included all randomized participants who received at least 1 infusion of PF-04360365. Here 'Number Analyzed' signifies participants evaluable for this measure at specified time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
units on a scale
  Baseline | 18.6 (8.71) | 23.5 (12.56) | 18.2 (6.57) | 20.1 (9.79)
  Change at Month 3: number analyzed (Participants) | 12 | 5 | 12 | 6
  Change at Month 3 | 0.5 (8.31) | 1.9 (5.43) | -2.6 (5.33) | -2.4 (3.72)
  Change at Month 6: number analyzed (Participants) | 12 | 6 | 12 | 5
  Change at Month 6 | 2.3 (5.96) | 2.3 (6.11) | -0.6 (7.32) | -4.3 (3.58)
  Change at Month 9: number analyzed (Participants) | 11 | 6 | 11 | 4
  Change at Month 9 | 2.4 (9.29) | 2.8 (11.00) | 1.6 (6.11) | -0.5 (6.34)
  Change at Month 13: number analyzed (Participants) | 10 | 4 | 11 | 3
  Change at Month 13 | 0.8 (6.27) | 0.9 (6.42) | 3.8 (8.04) | -2.0 (2.91)
  Change at Month 18: number analyzed (Participants) | 11 | 4 | 12 | 3
  Change at Month 18 | 5.4 (8.43) | -3.7 (0.72) | 5.9 (10.47) | 5.7 (5.51)
Statistical Analysis 1: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); Month 3: Mixed model repeated measures (MMRM) analysis with cohort, treatment by time interaction as fixed effects and baseline as covariate; Test type: Superiority or Other; p = 0.9779, Mixed Models Analysis; Least Squares (LS) Mean Difference = 0.11, 90% CI 2-sided [-6.49 to 6.71], Standard Error of Mean 3.959
Statistical Analysis 2: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); Month 6: Mixed model repeated measures (MMRM) analysis with cohort, treatment by time interaction as fixed effects and baseline as covariate; Test type: Superiority or Other; p = 0.8801, Mixed Models Analysis; LS Mean Difference = 0.58, 90% CI 2-sided [-5.79 to 6.94], Standard Error of Mean 3.815
Statistical Analysis 3: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); Month 9: Mixed model repeated measures (MMRM) analysis with cohort, treatment by time interaction as fixed effects and baseline as covariate; Test type: Superiority or Other; p = 0.9412, Mixed Models Analysis; LS Mean Difference = 0.28, 90% CI 2-sided [-6.13 to 6.70], Standard Error of Mean 3.845
Statistical Analysis 4: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); Month 13: Mixed model repeated measures (MMRM) analysis with cohort, treatment by time interaction as fixed effects and baseline as covariate; Test type: Superiority or Other; p = 0.7486, Mixed Models Analysis; LS Mean Difference = -1.36, 90% CI 2-sided [-8.38 to 5.66], Standard Error of Mean 4.223
Statistical Analysis 5: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); Month 18: Mixed model repeated measures (MMRM) analysis with cohort, treatment by time interaction as fixed effects and baseline as covariate; Test type: Superiority or Other; p = 0.0534, Mixed Models Analysis; L S Mean Difference = 8.18, 90% CI 2-sided [1.24 to 15.12], Standard Error of Mean 4.171
Statistical Analysis 6: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 1]; Test type: Superiority or Other; p = 0.9980, Mixed Models Analysis; L S Mean Difference = 0.01, 90% CI 2-sided [-6.29 to 6.31], Standard Error of Mean 3.776
Statistical Analysis 7: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 2]; Test type: Superiority or Other; p = 0.4004, Mixed Models Analysis; L S Mean Difference = 3.35, 90% CI 2-sided [-3.25 to 9.94], Standard Error of Mean 3.958
Statistical Analysis 8: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 3]; Test type: Superiority or Other; p = 0.6685, Mixed Models Analysis; L S Mean Difference = 1.81, 90% CI 2-sided [-5.20 to 8.82], Standard Error of Mean 4.214
Statistical Analysis 9: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 4]; Test type: Superiority or Other; p = 0.2968, Mixed Models Analysis; L S Mean Difference = 4.74, 90% CI 2-sided [-2.77 to 12.25], Standard Error of Mean 4.522
Statistical Analysis 10: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 5]; Test type: Superiority or Other; p = 0.7720, Mixed Models Analysis; L S Mean Difference = -1.31, 90% CI 2-sided [-8.77 to 6.16], Standard Error of Mean 4.494

52. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia (DAD) Total Score at Month 6, 13 and 18
Description: DAD is a functional assessment based on interview with the caregiver of participants. It consists of 40 items, 17 related to self-care and 23 items involving instrumental activities of daily living. Each item scored as yes = 1, no = 0 and not applicable= N/A. A total score is obtained by adding the rating for each question and converting this to a total score out of 100. The items rated N/A are not considered for the total score. DAD total score range from 0 (more dysfunction) to 100 (better function), with higher scores indicating better functioning.
Time Frame: Baseline, Month 6, 13, 18
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
units on a scale
  Baseline | 90.2 (12.58) | 85.6 (15.35) | 75.4 (17.85) | 87.3 (19.09)
  Change at Month 6 | -2.1 (4.51) | -3.4 (9.19) | -1.2 (13.06) | -1.0 (8.33)
  Change at Month 13: number analyzed (Participants) | 12 | 6 | 12 | 5
  Change at Month 13 | -9.5 (16.63) | -20.1 (22.81) | -8.5 (23.78) | -10.4 (19.10)
  Change at Month 18: number analyzed (Participants) | 12 | 6 | 11 | 5
  Change at Month 18 | -19.9 (21.43) | -28.0 (12.04) | -17.1 (24.18) | -14.7 (14.54)
Statistical Analysis 1: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); [analysis description as in outcome 51, analysis 2]; Test type: Superiority or Other; p = 0.8205, Mixed Models Analysis; LS Mean Difference = 2.00, 90% CI 2-sided [-12.68 to 16.69], Standard Error of Mean 8.789
Statistical Analysis 2: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); [analysis description as in outcome 51, analysis 4]; Test type: Superiority or Other; p = 0.2007, Mixed Models Analysis; LS Mean Difference = 11.37, 90% CI 2-sided [-3.31 to 26.06], Standard Error of Mean 8.789
Statistical Analysis 3: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); [analysis description as in outcome 51, analysis 5]; Test type: Superiority or Other; p = 0.3152, Mixed Models Analysis; LS Mean Difference = 8.90, 90% CI 2-sided [-5.78 to 23.59], Standard Error of Mean 0.8789
Statistical Analysis 4: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 2]; Test type: Superiority or Other; p = 0.8071, Mixed Models Analysis; LS Mean Difference = -2.20, 90% CI 2-sided [-17.18 to 12.79], Standard Error of Mean 8.964
Statistical Analysis 5: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 4]; Test type: Superiority or Other; p = 0.9918, Mixed Models Analysis; LS Mean Difference = -0.10, 90% CI 2-sided [-15.72 to 15.52], Standard Error of Mean 9.354
Statistical Analysis 6: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 51, analysis 5]; Test type: Superiority or Other; p = 0.7498, Mixed Models Analysis; LS Mean Difference = -3.01, 90% CI 2-sided [-18.73 to 12.70], Standard Error of Mean 9.415

53. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Total Score at Month 13
Description: Mini-Mental State Examination (MMSE) measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. Total MMSE score ranged from 0 (worst cognitive state) to 30 (best cognitive state), where higher score indicates better cognitive state.
Time Frame: Baseline, Month 13
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
units on a scale
  Baseline | 21.8 (3.81) | 20.3 (3.27) | 20.7 (3.68) | 21.7 (4.84)
  Change at Month 13: number analyzed (Participants) | 12 | 6 | 12 | 4
  Change at Month 13 | -1.5 (2.50) | -3.3 (6.68) | -1.3 (3.57) | -2.8 (3.20)
Statistical Analysis 1: Comparison: PF-04360365 10 mg/kg (Cohort Q) vs Placebo (Cohort Q); Month 13: Analysis of covariance (ANCOVA) with cohort by treatment interaction as fixed effect and baseline scores as covariate; Test type: Superiority or Other; p = 0.4855, ANCOVA; LS Mean Difference = 1.35, 90% CI 2-sided [-1.90 to 4.60], Standard Error of Mean 1.910
Statistical Analysis 2: Comparison: PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) vs Placebo (Cohort M); [analysis description as in outcome 53, analysis 1]; Test type: Superiority or Other; p = 0.5132, ANCOVA; LS Mean Difference = 1.45, 90% CI 2-sided [-2.27 to 5.16], Standard Error of Mean 2.185

54. Secondary Outcome: Mean Plasma Concentration of Amyloid Beta 1-x (A-beta 1-x)
Time Frame: Cohort M&Q: 0 hour(hr) & 0.25 hrs post dose (pd) on Day (D) 1,90,180,270,360, 0 hr pd on D 60,390; Cohort Q: 936,1176 hrs pd on D1(D 40,50); Cohort M: 216, 456 hrs pd on D1(D 10,20), 0.25 hrs pd on D 60, 0 hr & 0.25 hrs pd on D 30,120,150,210,240,300,330
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
pg/mL
  0 Hour Day 1 | 128.92 (129.49) | 136.00 (107.16) | 190.67 (133.79) | 167.17 (169.34)
  0.25 Hours Day 1: number analyzed (Participants) | 10 | 6 | 12 | 5
  0.25 Hours Day 1 | 454.50 (214.42) | 191.17 (97.01) | 551.33 (344.39) | 196.00 (152.32)
  0 Hour Day 10: number analyzed (Participants) | 0 | 0 | 4 | 1
  0 Hour Day 10 |  |  | 86025.00 (17717.48) | 171.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 20: number analyzed (Participants) | 0 | 0 | 3 | 2
  0 Hour Day 20 |  |  | 97633.33 (16223.54) | 268.50 (55.86)
  0 Hour Day 30: number analyzed (Participants) | 0 | 0 | 7 | 4
  0 Hour Day 30 |  |  | 112571.43 (20332.79) | 273.25 (125.07)
  0.25 Hours Day 30: number analyzed (Participants) | 0 | 0 | 5 | 4
  0.25 Hours Day 30 |  |  | 90900.00 (21793.12) | 288.25 (124.20)
  0 Hour Day 40: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 40 | 97225.00 (18871.56) | 266.00 (29.70) |  |
  0 Hour Day 50: number analyzed (Participants) | 3 | 2 | 0 | 0
  0 Hour Day 50 | 104833.33 (15671.10) | 299.00 (50.91) |  |
  0 Hour Day 60: number analyzed (Participants) | 3 | 2 | 6 | 3
  0 Hour Day 60 | 112100.00 (14255.88) | 455.50 (78.49) | 114650.00 (15162.55) | 234.33 (33.98)
  0.25 Hours Day 60: number analyzed (Participants) | 0 | 0 | 5 | 1
  0.25 Hours Day 60 |  |  | 115600.00 (8763.56) | 226.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 90: number analyzed (Participants) | 8 | 4 | 3 | 4
  0 Hour Day 90 | 69650.00 (19280.49) | 327.25 (162.98) | 107400.00 (14208.45) | 340.75 (183.38)
  0.25 Hours Day 90: number analyzed (Participants) | 8 | 4 | 3 | 4
  0.25 Hours Day 90 | 56450.00 (20203.96) | 349.50 (180.97) | 94166.67 (18315.11) | 381.00 (171.66)
  0 Hour Day 120: number analyzed (Participants) | 0 | 0 | 5 | 4
  0 Hour Day 120 |  |  | 114440.00 (20378.13) | 373.50 (181.21)
  0.25 Hours Day 120: number analyzed (Participants) | 0 | 0 | 4 | 1
  0.25 Hours Day 120 |  |  | 99425.00 (18753.38) | 249.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 150: number analyzed (Participants) | 0 | 0 | 5 | 3
  0 Hour Day 150 |  |  | 112920.00 (18388.37) | 276.67 (292.63)
  0.25 Hours Day 150: number analyzed (Participants) | 0 | 0 | 6 | 3
  0.25 Hours Day 150 |  |  | 100266.67 (28577.87) | 336.33 (233.34)
  0 Hour Day 180: number analyzed (Participants) | 3 | 1 | 6 | 3
  0 Hour Day 180 | 76533.33 (11019.23) | 459.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated. | 123333.33 (14066.51) | 280.33 (256.41)
  0.25 Hours Day 180: number analyzed (Participants) | 4 | 1 | 6 | 3
  0.25 Hours Day 180 | 67000.00 (12926.20) | 399.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated. | 106500.00 (20753.31) | 278.00 (297.64)
  0 Hour Day 210: number analyzed (Participants) | 0 | 0 | 5 | 3
  0 Hour Day 210 |  |  | 120400.00 (34173.09) | 265.33 (95.93)
  0.25 Hours Day 210: number analyzed (Participants) | 0 | 0 | 4 | 1
  0.25 Hours Day 210 |  |  | 103075.00 (18902.09) | 570.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 240: number analyzed (Participants) | 0 | 0 | 6 | 3
  0 Hour Day 240 |  |  | 115700.00 (22991.74) | 334.00 (430.61)
  0.25 Hours Day 240: number analyzed (Participants) | 0 | 0 | 5 | 3
  0.25 Hours Day 240 |  |  | 101700.00 (25123.69) | 303.33 (339.46)
  0 Hour Day 270: number analyzed (Participants) | 8 | 3 | 6 | 3
  0 Hour Day 270 | 72775.00 (16698.40) | 353.33 (127.41) | 114500.00 (10329.57) | 304.67 (358.70)
  0.25 Hours Day 270: number analyzed (Participants) | 1 | 3 | 6 | 2
  0.25 Hours Day 270 | 74000.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated. | 286.67 (105.04) | 104400.00 (23665.25) | 142.00 (200.82)
  0 Hour Day 300: number analyzed (Participants) | 0 | 0 | 4 | 3
  0 Hour Day 300 |  |  | 112750.00 (6075.91) | 230.67 (230.00)
  0.25 Hours Day 300: number analyzed (Participants) | 0 | 0 | 3 | 1
  0.25 Hours Day 300 |  |  | 101000.00 (19672.32) | 0.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 330: number analyzed (Participants) | 0 | 0 | 5 | 3
  0 Hour Day 330 |  |  | 119400.00 (31413.37) | 283.33 (251.46)
  0.25 Hours Day 330: number analyzed (Participants) | 0 | 0 | 4 | 3
  0.25 Hours Day 330 |  |  | 117000.00 (19899.75) | 256.33 (222.01)
  0 Hour Day 360: number analyzed (Participants) | 6 | 3 | 4 | 5
  0 Hour Day 360 | 81483.33 (11155.34) | 433.33 (128.94) | 115925.00 (21198.01) | 267.60 (188.12)
  0.25 Hours Day 360: number analyzed (Participants) | 8 | 0 | 5 | 5
  0.25 Hours Day 360 | 63462.50 (25395.10) |  | 111980.00 (19276.98) | 247.80 (226.73)
  0 Hour Day 390: number analyzed (Participants) | 0 | 2 | 1 | 0
  0 Hour Day 390 |  | 90.00 (127.28) | 140000.00 (NA) — Standard Deviation was not estimable since only 1 participant was evaluated. |

55. Secondary Outcome: Mean Plasma Concentration of Amyloid Beta 1-40 (A-beta 1-40)
Time Frame: Cohort M&Q: 0 hr & 0.25 hrs post dose(pd) on Day(D) 1,90,180,270,360, 0 hr pd on D 60,390,540; Cohort Q: 936, 1176 hrs pd on D1(D 40,50); Cohort M: 216, 456 hrs pd on D1(D 10,20), 0.25 hrs pd on D60, 0 hr & 0.25 hrs pd on D 30,120,150,210, 240,300,330
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
pg/mL
  0 Hour Day 1: number analyzed (Participants) | 9 | 5 | 10 | 5
  0 Hour Day 1 | 219.44 (163.52) | 136.60 (125.87) | 166.20 (102.44) | 157.20 (152.25)
  0.25 Hours Day 1: number analyzed (Participants) | 8 | 3 | 12 | 5
  0.25 Hours Day 1 | 618.00 (73.00) | 163.67 (141.99) | 530.33 (215.49) | 190.40 (26.29)
  0 Hour Day 10: number analyzed (Participants) | 0 | 0 | 3 | 0
  0 Hour Day 10 |  |  | 71233.33 (2345.92) |
  0 Hour Day 20: number analyzed (Participants) | 0 | 0 | 4 | 2
  0 Hour Day 20 |  |  | 97725.00 (29818.05) | 197.50 (28.99)
  0 Hour Day 30: number analyzed (Participants) | 0 | 0 | 11 | 6
  0 Hour Day 30 |  |  | 87045.45 (17785.41) | 216.00 (39.09)
  0.25 Hours Day 30: number analyzed (Participants) | 0 | 0 | 10 | 6
  0.25 Hours Day 30 |  |  | 93720.00 (14011.17) | 275.67 (120.27)
  0 Hour Day 40: number analyzed (Participants) | 3 | 0 | 0 | 0
  0 Hour Day 40 | 65100.00 (13163.97) |  |  |
  0 Hour Day 50: number analyzed (Participants) | 4 | 0 | 0 | 0
  0 Hour Day 50 | 105075.00 (26779.77) |  |  |
  0 Hour Day 60: number analyzed (Participants) | 4 | 2 | 12 | 6
  0 Hour Day 60 | 106625.00 (27207.15) | 269.50 (125.16) | 86383.33 (22189.79) | 137.67 (107.77)
  0.25 Hours Day 60: number analyzed (Participants) | 0 | 0 | 10 | 4
  0.25 Hours Day 60 |  |  | 91280.00 (25493.13) | 197.00 (133.61)
  0 Hour Day 90: number analyzed (Participants) | 9 | 3 | 12 | 6
  0 Hour Day 90 | 54244.44 (12650.31) | 225.67 (61.01) | 92341.67 (31491.97) | 179.17 (94.84)
  0.25 Hours Day 90: number analyzed (Participants) | 10 | 3 | 10 | 6
  0.25 Hours Day 90 | 50280.00 (15748.78) | 174.67 (163.48) | 73400.00 (29078.63) | 206.67 (74.95)
  0 Hour Day 120: number analyzed (Participants) | 0 | 0 | 12 | 6
  0 Hour Day 120 |  |  | 88850.00 (36003.07) | 243.83 (54.15)
  0.25 Hours Day 120: number analyzed (Participants) | 0 | 0 | 10 | 3
  0.25 Hours Day 120 |  |  | 78230.00 (32535.90) | 181.00 (158.09)
  0 Hour Day 150: number analyzed (Participants) | 0 | 0 | 9 | 5
  0 Hour Day 150 |  |  | 113788.89 (36944.09) | 1341.00 (1913.05)
  0.25 Hours Day 150: number analyzed (Participants) | 0 | 0 | 8 | 4
  0.25 Hours Day 150 |  |  | 107850.00 (44298.95) | 1422.00 (1655.19)
  0 Hour Day 180: number analyzed (Participants) | 12 | 6 | 7 | 6
  0 Hour Day 180 | 67566.67 (20145.35) | 228.17 (51.76) | 136800.00 (57309.80) | 623.50 (505.02)
  0.25 Hours Day 180: number analyzed (Participants) | 11 | 6 | 6 | 4
  0.25 Hours Day 180 | 62000.00 (20374.15) | 211.17 (107.37) | 154666.67 (67813.47) | 796.50 (502.64)
  0 Hour Day 210: number analyzed (Participants) | 0 | 0 | 7 | 2
  0 Hour Day 210 |  |  | 154142.86 (68875.32) | 696.50 (598.92)
  0.25 Hours Day 210: number analyzed (Participants) | 0 | 0 | 6 | 3
  0.25 Hours Day 210 |  |  | 139066.67 (62146.49) | 663.67 (413.37)
  0 Hour Day 240: number analyzed (Participants) | 0 | 0 | 7 | 4
  0 Hour Day 240 |  |  | 156714.29 (69257.28) | 616.25 (292.13)
  0.25 Hours Day 240: number analyzed (Participants) | 0 | 0 | 5 | 4
  0.25 Hours Day 240 |  |  | 128000.00 (43069.71) | 744.50 (533.68)
  0 Hour Day 270: number analyzed (Participants) | 8 | 6 | 6 | 3
  0 Hour Day 270 | 89062.50 (36384.45) | 607.17 (400.20) | 113766.67 (25223.53) | 473.67 (61.27)
  0.25 Hours Day 270: number analyzed (Participants) | 2 | 4 | 6 | 4
  0.25 Hours Day 270 | 95550.00 (43062.80) | 735.50 (481.31) | 150333.33 (43738.62) | 540.50 (382.69)
  0 Hour Day 300: number analyzed (Participants) | 0 | 0 | 6 | 6
  0 Hour Day 300 |  |  | 130000.00 (30880.41) | 607.50 (194.00)
  0.25 Hours Day 300: number analyzed (Participants) | 0 | 0 | 5 | 3
  0.25 Hours Day 300 |  |  | 138780.00 (72485.46) | 609.67 (204.23)
  0 Hour Day 330: number analyzed (Participants) | 0 | 0 | 7 | 5
  0 Hour Day 330 |  |  | 100285.71 (51435.12) | 1251.40 (1767.97)
  0.25 Hours Day 330: number analyzed (Participants) | 0 | 0 | 3 | 4
  0.25 Hours Day 330 |  |  | 103666.67 (81733.31) | 1545.75 (1545.67)
  0 Hour Day 360: number analyzed (Participants) | 7 | 6 | 8 | 3
  0 Hour Day 360 | 77442.86 (38989.14) | 1450.83 (2634.66) | 114612.50 (17519.82) | 1486.33 (1673.10)
  0.25 Hours Day 360: number analyzed (Participants) | 7 | 4 | 4 | 5
  0.25 Hours Day 360 | 70228.57 (33633.25) | 3287.50 (2585.41) | 131000.00 (33724.37) | 766.00 (685.10)
  0 Hour Day 390: number analyzed (Participants) | 0 | 3 | 0 | 2
  0 Hour Day 390 |  | 673.67 (629.67) |  | 330.00 (11.31)
  0 Hour Day 540: number analyzed (Participants) | 0 | 4 | 0 | 4
  0 Hour Day 540 |  | 369.00 (71.73) |  | 311.00 (37.26)

56. Secondary Outcome: Mean Plasma Concentration of Amyloid Beta 1-42 (A-beta 1-42)
Time Frame: Cohort M&Q: 0 hr & 0.25 hrs post dose(pd) on Day(D) 1,90,180,270,360, 0 hr pd on D 60,390; Cohort Q: 936, 1176 hrs pd on D1(D 40,50); Cohort M: 216, 456 hrs pd on D1(D 10,20), 0.25 hrs pd on D60, 0 hr & 0.25 hrs pd on D 30,120,150,210, 240,300,330
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
pg/mL
  0 Hour Day 1 | 4.62 (15.99) | 85.23 (133.09) | 41.05 (135.84) | 11.82 (28.94)
  0.25 Hours Day 1: number analyzed (Participants) | 10 | 6 | 12 | 5
  0.25 Hours Day 1 | 5.76 (18.21) | 73.23 (109.30) | 34.33 (112.18) | 15.96 (22.68)
  0 Hour Day 10: number analyzed (Participants) | 0 | 0 | 4 | 1
  0 Hour Day 10 |  |  | 0.00 (0.00) | 30.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 20: number analyzed (Participants) | 0 | 0 | 4 | 2
  0 Hour Day 20 |  |  | 141.25 (282.50) | 0.00 (0.00)
  0 Hour Day 30: number analyzed (Participants) | 0 | 0 | 11 | 6
  0 Hour Day 30 |  |  | 45.15 (139.88) | 17.48 (30.18)
  0.25 Hours Day 30: number analyzed (Participants) | 0 | 0 | 10 | 6
  0.25 Hours Day 30 |  |  | 47.24 (140.36) | 18.72 (33.96)
  0 Hour Day 40: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 40 | 0.00 (0.00) | 191.50 (270.82) |  |
  0 Hour Day 50: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 50 | 0.00 (0.00) | 46.15 (65.27) |  |
  0 Hour Day 60: number analyzed (Participants) | 4 | 2 | 12 | 6
  0 Hour Day 60 | 18.58 (37.15) | 0.00 (0.00) | 44.86 (135.13) | 17.43 (29.00)
  0.25 Hours Day 60: number analyzed (Participants) | 0 | 0 | 10 | 4
  0.25 Hours Day 60 |  |  | 37.12 (109.15) | 7.80 (15.60)
  0 Hour Day 90 | 6.18 (16.04) | 89.73 (138.77) | 43.19 (129.12) | 17.52 (31.33)
  0.25 Hours Day 90: number analyzed (Participants) | 11 | 6 | 10 | 6
  0.25 Hours Day 90 | 5.22 (17.31) | 87.67 (136.60) | 52.09 (152.20) | 14.77 (24.91)
  0 Hour Day 120: number analyzed (Participants) | 0 | 0 | 12 | 6
  0 Hour Day 120 |  |  | 45.19 (134.60) | 14.90 (25.03)
  0.25 Hours Day 120: number analyzed (Participants) | 0 | 0 | 10 | 3
  0.25 Hours Day 120 |  |  | 44.29 (124.45) | 17.40 (30.14)
  0 Hour Day 150: number analyzed (Participants) | 0 | 0 | 12 | 6
  0 Hour Day 150 |  |  | 42.48 (129.48) | 4.28 (10.49)
  0.25 Hours Day 150: number analyzed (Participants) | 0 | 0 | 11 | 6
  0.25 Hours Day 150 |  |  | 45.51 (132.38) | 4.67 (11.43)
  0 Hour Day 180 | 6.52 (15.24) | 77.83 (131.64) | 16.67 (57.74) | 0.00 (0.00)
  0.25 Hours Day 180: number analyzed (Participants) | 11 | 6 | 10 | 6
  0.25 Hours Day 180 | 3.69 (12.24) | 78.83 (124.29) | 14.70 (46.49) | 0.00 (0.00)
  0 Hour Day 210: number analyzed (Participants) | 0 | 0 | 12 | 5
  0 Hour Day 210 |  |  | 3.96 (13.71) | 0.00 (0.00)
  0.25 Hours Day 210: number analyzed (Participants) | 0 | 0 | 12 | 3
  0.25 Hours Day 210 |  |  | 21.08 (73.03) | 0.00 (0.00)
  0 Hour Day 240: number analyzed (Participants) | 0 | 0 | 12 | 5
  0 Hour Day 240 |  |  | 3.18 (11.00) | 0.00 (0.00)
  0.25 Hours Day 240: number analyzed (Participants) | 0 | 0 | 11 | 5
  0.25 Hours Day 240 |  |  | 38.73 (128.44) | 0.00 (0.00)
  0 Hour Day 270: number analyzed (Participants) | 11 | 6 | 12 | 5
  0 Hour Day 270 | 0.00 (0.00) | 96.83 (168.84) | 22.50 (77.94) | 0.00 (0.00)
  0.25 Hours Day 270: number analyzed (Participants) | 7 | 6 | 11 | 4
  0.25 Hours Day 270 | 0.00 (0.00) | 79.33 (141.85) | 1.85 (6.15) | 0.00 (0.00)
  0 Hour Day 300: number analyzed (Participants) | 0 | 0 | 11 | 6
  0 Hour Day 300 |  |  | 38.91 (129.05) | 0.00 (0.00)
  0.25 Hours Day 300: number analyzed (Participants) | 0 | 0 | 10 | 3
  0.25 Hours Day 300 |  |  | 14.60 (46.17) | 0.00 (0.00)
  0 Hour Day 330: number analyzed (Participants) | 0 | 0 | 12 | 5
  0 Hour Day 330 |  |  | 0.00 (0.00) | 0.00 (0.00)
  0.25 Hours Day 330: number analyzed (Participants) | 0 | 0 | 10 | 5
  0.25 Hours Day 330 |  |  | 0.00 (0.00) | 0.00 (0.00)
  0 Hour Day 360: number analyzed (Participants) | 12 | 6 | 12 | 5
  0 Hour Day 360 | 0.00 (0.00) | 98.33 (165.43) | 44.59 (146.44) | 0.00 (0.00)
  0.25 Hours Day 360: number analyzed (Participants) | 11 | 6 | 11 | 5
  0.25 Hours Day 360 | 0.00 (0.00) | 130.17 (265.68) | 31.64 (104.93) | 0.00 (0.00)
  0 Hour Day 390: number analyzed (Participants) | 9 | 5 | 12 | 4
  0 Hour Day 390 | 0.00 (0.00) | 107.40 (240.15) | 12.17 (42.15) | 0.00 (0.00)

57. Other Pre Specified Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Total Tau and Phospho-tau (P-tau) Proteins
Time Frame: Cohort M&Q: Pre dose (0 hr) on Day 0, 0 hr post dose on Day 180, 360; Cohort Q: 936, 1176 hrs post dose on Day 1(Day 40,50), 0 hr post dose on Day 60, 90; Cohort M: 216, 456 hrs post dose on Day 1(Day 10, 20), 0 hr post dose on Day 30
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
pg/mL
  0 Hour Day 0: tau | 185.70 (58.11) | 194.00 (88.75) | 140.93 (50.96) | 165.83 (49.77)
  0 Hour Day 10: tau: number analyzed (Participants) | 0 | 0 | 4 | 1
  0 Hour Day 10: tau |  |  | -15.09 (16.44) | 2.55 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 20: tau: number analyzed (Participants) | 0 | 0 | 4 | 1
  0 Hour Day 20: tau |  |  | -11.67 (12.82) | 4.72 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 30: tau: number analyzed (Participants) | 0 | 0 | 4 | 2
  0 Hour Day 30: tau |  |  | 6.60 (17.76) | 4.22 (1.36)
  0 Hour Day 40: tau: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 40: tau | -21.13 (9.99) | -4.07 (3.13) |  |
  0 Hour Day 50: tau: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 50: tau | 7.70 (24.02) | 7.92 (6.19) |  |
  0 Hour Day 60: tau: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 60: tau | 15.90 (22.71) | -10.43 (3.35) |  |
  0 Hour Day 90: tau: number analyzed (Participants) | 4 | 1 | 0 | 0
  0 Hour Day 90: tau | -6.88 (22.64) | -9.18 (NA) — Standard deviation was not estimable since only 1 participant was evaluated. |  |
  0 Hour Day 180: tau: number analyzed (Participants) | 8 | 4 | 11 | 4
  0 Hour Day 180: tau | -15.76 (18.49) | -37.35 (13.67) | -16.47 (22.01) | 8.60 (7.16)
  0 Hour Day 360: tau: number analyzed (Participants) | 10 | 6 | 11 | 4
  0 Hour Day 360: tau | 1.37 (22.13) | -2.07 (19.78) | -13.15 (21.38) | -9.75 (9.61)
  0 Hour Day 0: p-tau | 67.19 (18.05) | 65.77 (20.21) | 60.27 (26.26) | 74.00 (27.73)
  0 Hour Day 10: p-tau: number analyzed (Participants) | 0 | 0 | 4 | 1
  0 Hour Day 10: p-tau |  |  | 0.25 (36.71) | 32.52 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 20: p-tau: number analyzed (Participants) | 0 | 0 | 4 | 1
  0 Hour Day 20: p-tau |  |  | 24.79 (73.39) | 34.55 (NA) — Standard deviation was not estimable since only 1 participant was evaluated.
  0 Hour Day 30: p-tau: number analyzed (Participants) | 0 | 0 | 4 | 2
  0 Hour Day 30: p-tau |  |  | 2.91 (6.51) | 0.92 (3.82)
  0 Hour Day 40: p-tau: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 40: p-tau | 21.41 (27.96) | 6.53 (1.72) |  |
  0 Hour Day 50: p-tau: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 50: p-tau | 39.51 (63.57) | 62.96 (100.89) |  |
  0 Hour Day 60: p-tau: number analyzed (Participants) | 4 | 2 | 0 | 0
  0 Hour Day 60: p-tau | 2.28 (19.79) | -3.10 (10.26) |  |
  0 Hour Day 90: p-tau: number analyzed (Participants) | 4 | 1 | 0 | 0
  0 Hour Day 90: p-tau | 16.04 (24.13) | -3.95 (NA) — Standard deviation was not estimable since only 1 participant was evaluated. |  |
  0 Hour Day 180: p-tau: number analyzed (Participants) | 8 | 4 | 12 | 5
  0 Hour Day 180: p-tau | -8.31 (29.96) | -7.45 (43.56) | -10.79 (58.37) | 10.04 (24.97)
  0 Hour Day 360: p-tau: number analyzed (Participants) | 12 | 6 | 12 | 4
  0 Hour Day 360: p-tau | 4.29 (38.32) | 24.55 (35.01) | 8.96 (68.60) | -7.31 (41.09)

58. Other Pre Specified Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Protein Concentration at Day 10, 20, 30, 40, 50, 60, 90, 180 and 360
Time Frame: Cohort M&Q: Baseline, 0 hr post dose on Day 180, 360; Cohort Q: 936, 1176 hrs post dose on Day 1(Day 40,50), 0 hr post dose on Day 60, 90; Cohort M: 216, 456 hrs post dose on Day 1(Day 10, 20), 0 hr post dose on Day 30
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
gram per liter (g/L)
  Baseline | 0.32 (0.091) | 0.30 (0.230) | 0.32 (0.198) | 0.22 (0.050)
  Change at 0 Hour Day 10: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 10 |  |  | -0.01 (0.013) | 0.01 (0.011)
  Change at 0 Hour Day 20: number analyzed (Participants) | 0 | 0 | 4 | 1
  Change at 0 Hour Day 20 |  |  | 0.04 (0.077) | 0.01 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at 0 Hour Day 30: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 30 |  |  | 0.02 (0.027) | 0.00 (0.014)
  Change at 0 Hour Day 40: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 40 | 0.00 (0.015) | 0.02 (0.013) |  |
  Change at 0 Hour Day 50: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 50 | 0.00 (0.031) | 0.06 (0.064) |  |
  Change at 0 Hour Day 60: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 60 | 0.02 (0.108) | 0.07 (0.080) |  |
  Change at 0 Hour Day 90: number analyzed (Participants) | 4 | 1 | 0 | 0
  Change at 0 Hour Day 90 | -0.01 (0.015) | 0.01 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |
  Change at 0 Hour Day 180: number analyzed (Participants) | 8 | 4 | 12 | 5
  Change at 0 Hour Day 180 | 0.04 (0.088) | 0.09 (0.081) | 0.02 (0.029) | 0.04 (0.026)
  Change at 0 Hour Day 360: number analyzed (Participants) | 12 | 6 | 12 | 5
  Change at 0 Hour Day 360 | 0.02 (0.059) | 0.05 (0.056) | 0.00 (0.036) | 0.02 (0.017)

59. Other Pre Specified Outcome: Change From Baseline in Red Blood Cells (RBCs) and White Blood Cells (WBCs) Concentration in Cerebrospinal Fluid (CSF) at Day 10, 20, 30, 40, 50, 60, 90, 180, 360
Time Frame: as for outcome 58
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: 10^6 cells per liter
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
10^6 cells per liter
  Baseline: RBC | 30.08 (83.842) | 1.17 (2.041) | 2.58 (2.392) | 8.17 (12.287)
  Change at 0 Hour Day 10: RBC: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 10: RBC |  |  | -0.25 (0.500) | 67.50 (95.459)
  Change at 0 Hour Day 20: RBC: number analyzed (Participants) | 0 | 0 | 4 | 1
  Change at 0 Hour Day 20: RBC |  |  | 80.50 (141.576) | -18.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at 0 Hour Day 30: RBC: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 30: RBC |  |  | 12.75 (25.513) | 1.50 (2.121)
  Change at 0 Hour Day 40: RBC: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 40: RBC | -75.75 (146.227) | 0.50 (0.707) |  |
  Change at 0 Hour Day 50: RBC: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 50: RBC | -4.50 (9.000) | 0.00 (0.000) |  |
  Change at 0 Hour Day 60: RBC: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 60: RBC | 2.50 (8.660) | 0.00 (0.000) |  |
  Change at 0 Hour Day 90: RBC: number analyzed (Participants) | 4 | 1 | 0 | 0
  Change at 0 Hour Day 90: RBC | -70.75 (149.295) | -1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |
  Change at 0 Hour Day 180: RBC: number analyzed (Participants) | 8 | 4 | 12 | 5
  Change at 0 Hour Day 180: RBC | 72.00 (191.426) | 1.75 (2.217) | 6.25 (15.516) | 24.60 (62.528)
  Change at 0 Hour Day 360: RBC: number analyzed (Participants) | 12 | 6 | 12 | 5
  Change at 0 Hour Day 360: RBC | -26.67 (84.610) | 21.83 (37.870) | 26.67 (74.644) | -6.80 (9.960)
  Baseline: WBC | 1.34 (1.310) | 0.98 (1.250) | 1.47 (1.798) | 1.42 (1.563)
  Change at 0 Hour Day 10: WBC: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 10: WBC |  |  | 0.50 (2.517) | 0.00 (0.000)
  Change at 0 Hour Day 20: WBC: number analyzed (Participants) | 0 | 0 | 4 | 1
  Change at 0 Hour Day 20: WBC |  |  | 0.50 (1.000) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at 0 Hour Day 30: WBC: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 30: WBC |  |  | 0.00 (0.000) | -0.30 (0.424)
  Change at 0 Hour Day 40: WBC: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 40: WBC | 0.75 (0.957) | -0.50 (0.707) |  |
  Change at 0 Hour Day 50: WBC: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 50: WBC | 0.35 (1.814) | -0.65 (0.919) |  |
  Change at 0 Hour Day 60: WBC: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 60: WBC | -0.48 (0.618) | 0.30 (0.424) |  |
  Change at 0 Hour Day 90: WBC: number analyzed (Participants) | 4 | 1 | 0 | 0
  Change at 0 Hour Day 90: WBC | 1.00 (1.155) | -1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |
  Change at 0 Hour Day 180: WBC: number analyzed (Participants) | 8 | 4 | 12 | 5
  Change at 0 Hour Day 180: WBC | -0.35 (0.862) | -0.33 (1.087) | 0.06 (0.876) | 0.14 (0.699)
  Change at 0 Hour Day 360: WBC: number analyzed (Participants) | 12 | 6 | 12 | 5
  Change at 0 Hour Day 360: WBC | -0.04 (2.097) | -0.48 (0.801) | 0.22 (0.944) | 0.14 (1.182)

60. Other Pre Specified Outcome: Change From Baseline in Glucose Concentration in Cerebrospinal Fluid (CSF) at Day 10, 20, 30, 40, 50, 60, 90, 180, 360
Time Frame: as for outcome 58
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Number analyzed (Participants) | 12 | 6 | 12 | 6
millimole per liter (mmol/L)
  Baseline | 3.47 (0.267) | 3.40 (0.438) | 3.41 (0.188) | 3.35 (0.288)
  Change at 0 Hour Day 10: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 10 |  |  | 0.00 (0.082) | -0.20 (0.141)
  Change at 0 Hour Day 20: number analyzed (Participants) | 0 | 0 | 4 | 1
  Change at 0 Hour Day 20 |  |  | 0.03 (0.126) | -0.10 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at 0 Hour Day 30: number analyzed (Participants) | 0 | 0 | 4 | 2
  Change at 0 Hour Day 30 |  |  | -0.03 (0.206) | 0.00 (0.141)
  Change at 0 Hour Day 40: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 40 | -0.10 (0.141) | 0.10 (0.283) |  |
  Change at 0 Hour Day 50: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 50 | -0.08 (0.171) | 0.05 (0.071) |  |
  Change at 0 Hour Day 60: number analyzed (Participants) | 4 | 2 | 0 | 0
  Change at 0 Hour Day 60 | -0.08 (0.275) | -0.30 (0.283) |  |
  Change at 0 Hour Day 90: number analyzed (Participants) | 4 | 1 | 0 | 0
  Change at 0 Hour Day 90 | 0.00 (0.216) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |
  Change at 0 Hour Day 180: number analyzed (Participants) | 8 | 4 | 12 | 5
  Change at 0 Hour Day 180 | -0.01 (0.295) | -0.18 (0.411) | -0.01 (0.156) | 0.00 (0.187)
  Change at 0 Hour Day 360: number analyzed (Participants) | 12 | 6 | 12 | 5
  Change at 0 Hour Day 360 | -0.03 (0.246) | 0.00 (0.358) | 0.58 (1.012) | 0.04 (0.182)

61. Other Pre Specified Outcome: Number of Participants With Measurable Serum Anti-Drug Antibody (ADA) Concentration
Description: A measurable ADA is defined as a serum anti-drug anti body response (total binding assay) greater than the lower limit of quantification (4.32).
Time Frame: Day 1 up to Month 18
Population: Safety analysis set included all randomized participants who received at least 1 infusion of PF-04360365. Only participants receiving PF-04360365 were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study. Data for adverse events were summarized by cohort as pre-specified in statistical analysis plan; hence, combined data is presented for PF-04360365 10 mg/kg, then PF-04360365 7.5 mg/kg (Cohort M).
Arm/Group | PF-04360365 10 mg/kg (Cohort Q) | Placebo (Cohort Q) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) | Placebo (Cohort M)
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/6 | 1/12 | 0/6
Other Adverse Events (participants affected / at risk) | 9/12 | 5/6 | 10/12 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04360365 10 mg/kg (Cohort Q) (N=12) | Placebo (Cohort Q) (N=6) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) (N=12) | Placebo (Cohort M) (N=6)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04360365 10 mg/kg (Cohort Q) (N=12) | Placebo (Cohort Q) (N=6) | PF-04360365 10 mg/kg, Then PF-04360365 7.5 mg/kg (Cohort M) (N=12) | Placebo (Cohort M) (N=6)
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Tenderness (General disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Areflexia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 4 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.